CLINICAL TRIAL: NCT05536934
Title: Arginase Inhibition and Endothelial Function in Humans With Obesity
Brief Title: Arginase Inhibition in Humans With Obesity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, John Pernow, Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016/1173-32
Record Dates: First submitted 2022-08-21; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Obese; Endothelial Function
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arginase inhibition (Experimental): Endothelium dependent and -independent vasodilatation before and after 120min intra-arterial administration of arginase the inhibitor N-omega-hydroxy-nor-l-arginine (nor-NOHA) is started and is maintained for 120 min at a rate of 0.1 mg/min
  Interventions: Drug: Nω-hydroxy-nor-arginine

INTERVENTIONS:
Drug: Nω-hydroxy-nor-arginine

SUMMARY:
To evaluate the efficacy of arginase inhibition on endothelial function in humans with obesity.

DETAILED DESCRIPTION:
The study is performed on one group of subjects with body mass index >35 and the absence of type 2 diabetes.

Inclusion criteria:

Body mass index >35 kg/m2.

Exclusion criteria:

Age >80 years. Type 2 diabetes defined as >7 mmol/L in fasting plasma glucose or >11 mmol/L following 2h of oral glycemic load.

Myocardial infarction/unstable angina within 6 weeks prior to the study. Treatment with oral anticoagulants (Warfarin or New oral anticoagulants), Raynaud's phenomenon, peripheral vasculopathies, arterial shunting or other vascular surgery of the study arm.

Any concomitant disease or condition that may interfere with the possibility for the patient to comply with or complete the study protocol.

Participant in an ongoing study. Unwillingness to participate following oral and written information.

Forearm blood flow is determined by venous occlusion plethysmography. Endothelium-dependent vasodilatation is determined during intra-brachial artery infusion of serotonin (21, 70 and 210 ng/min). Endothelium-independent vasodilatation is determined by infusion of sodium nitroprusside (SNP; 1, 3 and 10 µg/min). Each dose is given for 2 min at a rate of 2.5 ml/min. Data are expressed as percentage change in forearm blood from baseline flow.

Fifteen subjects are included. On the day of the study the subject arrives to the laboratory after having a light breakfast. Forearm vessels of the non-dominant arm are cannulated and forearm blood flow is determined as described above. Baseline endothelium-dependent and endothelium-independent vasodilatation is determined by intra-arterial infusions of serotonin and SNP, respectively. Thereafter an intra-arterial infusion of the arginase inhibitor N-omega-hydroxy-nor-l-arginine (nor-NOHA) is administered as an intra-arterial infusion at a rate of 0.1 mg/min and is maintained for 120 min. The dose is based on a previous study by our group demonstrating improved endothelial function. Endothelium-dependent and -independent vasodilatation is reassessed at 120 min of infusion.

ELIGIBILITY:
Inclusion Criteria:

BMI >35kg/m2

Exclusion Criteria:

Age >80 years. Type 2 diabetes defined as >7 mmol/L in fasting plasma glucose or >11 mmol/L following 2h of oral glycemic load.

Myocardial infarction/unstable angina within 6 weeks prior to the study. Treatment with oral anticoagulants (Warfarin or New oral anticoagulants), Raynaud's phenomenon, peripheral vasculopathies, arterial shunting or other vascular surgery of the study arm.

Any concomitant disease or condition that may interfere with the possibility for the patient to comply with or complete the study protocol.

Participant in an ongoing study. Unwillingness to participate following oral and written information.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Endothelium-dependent change in forearm blood flow | 120 min intraarterial infusion of the arginase inhibitor nor-NOHA
  Percentage change in forearm blood flow from baseline induced by the endothelium-dependent vasodilator serotonin during arginase blockade vs. saline.

SECONDARY OUTCOMES:
Endothelium-independent change in forearm blood flow | 120 min intraarterial infusion of the arginase inhibitor nor-NOHA
  Percentage change in forearm blood flow from baseline induced by the endothelium-independent vasodilator nitroprusside during arginase blockade vs. saline.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No